CLINICAL TRIAL: NCT04499040
Title: Tricho-hepato-enteric Syndrome: From Abnormal RNA Decay to Disease Clinical and Biological Characterization of Patients and Collection of Samples -THE-RNA
Brief Title: Clinical and Biological Characterization of Patients and Collection of Samples
Acronym: THE-RNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-42
Record Dates: First submitted 2016-08-31; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Tricho Hepato Enteric Syndrome
MeSH Terms: conditions — Trichohepatoenteric Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with SD/THE (Experimental)
  Interventions: Biological: Blood sample; Other: Fecal samples; Behavioral: Neuropsychological
- control group (Placebo Comparator)
  Interventions: Biological: Blood sample; Other: Fecal samples

INTERVENTIONS:
Biological: Blood sample — Blood samples to assess biological parameters such as:
Other: Fecal samples — Microbiota analysis
Behavioral: Neuropsychological — Neuropsychological assessment
  Arms: patients with SD/THE

SUMMARY:
Objectives: Collect clinical and biological data about patients with SD/THE, collect samples of patients; create a secure on line database to collect worldwide data about SD/THE Partners : APHM, HCL, APHP

Currently10 patients (8 with TTC37 mutations and 2 with SKIV2l mutations) present a SD/THE and are managed in France in 5 different centers (Marseille, Paris Trousseau, Paris Necker, Paris Robert Debrés, and Lyon). Most of them are followed in hepato-gastro-enterology units for their intractable diarrhea. Three aspects of the disease: intractable diarrhea, immune defect and liver disease are responsible for the main part of the burden of the disease .For each aspect, the investigators will propose a close follow-up with collection of clinical, biochemical, functional and microbial data.

Collect of clinical date: during a programmed consultation clinical data about symptom will be collected twice a year. A detailed form will be used for better delineation of the symptoms. These data included growth, symptom (diarrhea, pain …), and clinical signs. Most of these children have recurrent sample for follow up. During them some blood will be take for study the immune side but also the platelet function.

ELIGIBILITY:
Inclusion Criteria:

* patient < 18 year-old
* patients with SD/THE

control group :

* patients with tufting enteropathy and short bowel syndrome.

Exclusion Criteria:

* child among whom the parents or the legal representatives refused that their child participates in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of detailed clinical characteristics of the phenotype of Tricho-hepato-enteric syndrome | 3 years
  Existence or absence of 9 clinical signs suggestive of Tricho-hepato-enteric syndrome, to know:
  * neonatal characteristics,
  * existence or not of the 9 clinical signs suggestive of the disease,
  * initial symptoms and chronology leading to the diagnosis,
  * organ damage,
  * nutrition,
  * treatment,
  * growth,
  * dermatological evaluation,
  * hepatic evaluation,
  * neuropsychological evaluation (score of WPPSI-III, WISC-IV, WAIS-IV),
  * quality of life scale (VSPA in children between 3 and 17 years old and WHOQUOL in adults),
  * self-report anxiety scale (STAI in children over 8 years)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier Arnaud, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No